CLINICAL TRIAL: NCT07021183
Title: Uptake, Acceptability, and Effectiveness of Internet-Delivered Cognitive Behaviour Therapy for Public Safety Personnel With Self-Reported Sleep Difficulties
Brief Title: The Public Safety Personnel (PSP) Sleep Course: An Online Sleep Intervention for PSP.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Collaborators: Government of Canada (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1088
Record Dates: First submitted 2025-03-31; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2024-12

CONDITIONS: Insomnia
Keywords: Internet; Internet-Delivered CBT; Digital Mental Health Interventions; Insomnia; Sleep Difficulties; Depression; Anxiety; Public Safety Personnel
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ICBT for insomnia (Experimental): Therapist-guided, internet-delivered cognitive behavioral therapy for insomnia (ICBTi)
  Interventions: Behavioral: Sleep Course

INTERVENTIONS:
Behavioral: Sleep Course — The Sleep Course previously developed and evaluated in Australia will be delivered to clients meeting participation criteria tailored to PSP. The Sleep Course has been slightly adapted for PSP by including relevant statistics and literature pertaining to sleep disturbance in PSP. The Sleep Course has four lessons and includes optional therapist support for up to 8 - 12 weeks. Should clients request support, clients will be contacted by their therapist by secure emails on their designated check-in dates. The therapist also reviews client progress in the Course and emails clients on a designated check in date. Sometimes the therapist will call the client. Phone calls are typically made if a client is not logging in or if the therapist feels that a phone call would be a helpful way to provide support.

SUMMARY:
This study evaluates an internet-delivered cognitive behavioural therapy for insomnia (ICBTi) intervention, known as the Sleep Course, adapted for public safety personnel (PSP) experiencing sleep difficulties. The study seeks to replicate prior results from an Australian version of the Sleep Course assessing its effectiveness and acceptability when offered to PSP.

DETAILED DESCRIPTION:
Background:

Public safety personnel (PSP) refer to individuals who ensure the safety and security of their citizens (e.g., border services officers, correctional workers, firefighters, paramedics, police). These occupations often require long and irregular hours (e.g., shift work) which can negatively impact daily functioning and work performance. PSP also experience increased exposure to potentially psychologically traumatic events (PPTEs) which can increase risk for mental health challenges (e.g., anxiety, depression, posttraumatic stress). These occupational stressors can also lead to sleep disturbance among PSP. Contributing factors to PSP sleep difficulties include long work hours, varying shift work, high stress, and exposure to PPTEs. Some evidence suggests that certain sectors are more susceptible to sleep difficulties, with correctional workers, paramedics, and Royal Canadian Mounted Police (RCMP) more difficulties than firefighters and police officers.

To improve access to effective psychological treatment, internet-delivered cognitive behaviour therapy (ICBT) has emerged as a structured online alternative to face-to-face cognitive behaviour therapy (CBT) in which treatment materials are delivered periodically over several months. The approach can be offered with or without therapist support. Research supports the effectiveness of ICBT for conditions like depression, anxiety, alcohol misuse, and insomnia with outcomes comparable to face-to-face therapy. Moreover, there is evidence that PSP benefit from transdiagnostic and PTSD-specific ICBT but to date there are no studies exploring ICBTi among PSP.

Individuals who experience sleep disturbances are more likely to report increased physical (e.g., illness, poor health, pain) and mental challenges (e.g., anxiety, depression), as well as decreased work performance, daily functioning, and quality of life. PSP similarly experience these effects of sleep disturbances.

Internet-delivered cognitive behaviour therapy for insomnia (ICBTi) is an evidence-based treatment for insomnia and sleep diﬃculties. Studying this among PSP is important as access to specialized psychological services, such as CBTi, is often limited, even though CBTi is a well-established treatment, and generally preferred over medication. ICBTi offers a promising approach for expanding access to evidence-based treatment for insomnia. The current study aims to explore the extent to which this ICBTi program, called the Sleep Course will be used by PSP, found to be acceptable and effective. Findings will shape long-term practices of working with PSP, contribute to a broader understanding of how ICBTi can address insomnia in PSP, and address the personal and societal impacts of untreated insomnia.

Research purpose:

The purpose of this research project is to offer and evaluate an ICBTi program, the Sleep Course, for PSP. Key objectives are to examine: 1) the uptake and completion rates of the Sleep Course among PSP, 2) the baseline demographic and clinical characteristics of PSP enrolled in the program, 3) clients' acceptability ratings and feedback, 4) reductions in sleep-related measures, and 5) reductions in secondary measures.

To take part in this study, PSP will undergo a two-stage intake process: First, interested individuals will complete an online screening questionnaire that assesses a variety of clinical characteristics pre-treatment. Second, participants who meet initial inclusion criteria will be enrolled in the program and matched with a clinician. Those who do not meet initial inclusion criteria will be given the option of scheduling a phone interview with a clinician to further discuss their eligibility.

All clients will receive the same Sleep Course, which was developed at Macquarie University, Australia. The Sleep Course is an intervention targeting sleep concerns. It comprises 4 online lessons that provide: 1) psychoeducation on sleep (week 1); 2) information on sleep restriction and stimulus control strategies (week 2); 3) information on thought monitoring and challenging and worry time (week 4); and 4) behavioural strategies including activity scheduling and wind down and up routines (week 6). Lessons will be released gradually in a standardized order over 6 weeks with regular automatic emails informing clients about upcoming lessons. Supplementary resources can be accessed at any time but are recommended as follows: Lesson 1 Myth-busting; Lesson 2 Shift Work, Diet, Medication & Exercise; Lesson 3 Relaxation and Nightmares; and Lesson 4 Maintaining Progress. Materials are presented in a didactic (i.e., text-based with visual images) and case-enhanced learning format (i.e., educational stories demonstrate the application of skills). Each of the 4 lessons offers Do-It-Yourself Exercises that facilitate skill acquisition for all clients.

Once enrolled in the Sleep Course, clients will be able to email their assigned therapist at any time for 8 weeks, with the possibility of extending care up to 12 weeks. Should they request support clients will be contacted by their therapist by secure emails on their designated check-in dates. Therapists will offer support and encouragement related to the Sleep Course content and answer any client questions. Therapists will also contact clients by phone if therapists are concerned about client safety, if clients have not logged in to the Sleep Course, or if clients request a phone call instead of email.

The primary research questions to be answered are:

1. What will be the uptake and completion of the Sleep Course among PSP?
2. What are the baseline demographic and clinical characteristics of PSP who are enrolled in the Sleep Course?
3. How acceptable is the Sleep Course as assessed via participants' ratings and feedback?
4. Will the Sleep Course result in significant reductions on sleep-related and secondary measures?

Significance:

The data collected will shape long-term practices within our unit that provides ICBT to PSP and has potential to significantly enhance service delivery. The research will also provide valuable insights for other online clinics regarding the potential of offering ICBTi to PSP. By exploring the program's use, client characteristics, acceptability, and effectiveness, this study will contribute to a broader understanding of how ICBTi can be offered to PSP ultimately improving access to evidence-based treatment for insomnia.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of older
* Current or former paid or volunteer PSP
* Living in a province in Canada where we offer the PSP Sleep Couse for the treatment period
* Willingness to learn information and skills to self-manage sleep difficulties
* Have internet access
* Consent to Sleep Course, online therapy as provided by PSPNET, and associated research

Exclusion Criteria:

* Current severe medical or psychiatric disorder (e.g. current and recent mania or psychosis, recent hospitalization for mental health concerns, actively suicidal, medical condition client thinks will interfere with treatment, severe substance use)
* Unable to read and understand English. (All content is provided in English and staﬀ is English speaking; pending findings of the research we will explore translating the course into French)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in insomnia | Screening, week 7 (post-treatment), and 3-month follow-up
  Insomnia Severity Index (ISI). Includes 7 items rated on a 0 to 5 scale. Higher total scores indicate greater severity of insomnia symptoms over the past two weeks. Scores range from 0 to 28.

SECONDARY OUTCOMES:
Change in Sleep Quality | Screening, start of lesson 1 (day 0), start of lesson 2 (day 7), start of lesson 3 (day 21), start of lesson 4 (day 35), and week 7 (post-treatment), and 3-month follow-up
  Sleep Quality Scale (SQS) is a 1-item survey that assess overall sleep quality for over the past week.
Change in Sleep-Related Impairment | Screening, week 7 (post-treatment), and 3 month follow up
  The PROMIS Sleep Related Impairment Short Form (SRI-SF) scale assesses the impact of sleep disturbances on daytime functioning. There are 8 items, which are related to cognitive, emotional, and social functioning. Responses range from 0 (not at all) to 4 (very much).
Change in attitudes and beliefs about sleep | Screening, week 7 (post-treatment) and 3-month follow-up
  Dysfunctional Beliefs and Attitudes about Sleep- 16 item (DBAS-16) with items rated on a 0 to 10-point scale. Scores range from 0 to 160 with higher scores indicating greater dysfunctional beliefs about sleep.
Change in depression | Screening, week 7 (post-treatment) and 3-month follow-up
  Patient Health Questionnaire - 9 Item (PHQ-9). Includes 9 items rated 0 to 3. Higher total scores indicate greater severity of depression. Scores range from 0 to 27. Clinical cutoff of ≥10 indicate clinically significant depression.
Change in anxiety | Screening, week 7 (post treatment) and 3-month follow-up
  Generalized Anxiety Disorder - 7 Item (GAD-7). Includes 7 items rated 0 to 3. Higher total scores indicate greater severity of anxiety. Scores range from 0 to 21. Clinical cutoff of ≥10 indicates clinically significant anxiety.
Change in posttraumatic stress | Screening, week 7 (post treatment) and 3-month follow-up
  Abbreviated PTSD Checklist - Civilian Version (PCL-C). Six items. Higher total scores indicate greater severity of posttraumatic stress. Scores range from 5 to 30.
Lesson reflection | At the end of Lesson 1 (day 0), Lesson 2 (day 7), Lesson 3 (day 21), and Lesson 4 (day 35).
  Lesson reflection questionnaire - A bespoke 5-item survey that inquires about how understandable and helpful the lesson was, client successes or challenges over the previous week, and suggestions for improvement. This survey is used for clinicians to monitor treatment. No overall score is created.
Evaluation of treatment | Week 7 (post-treatment)
  Treatment Satisfaction Survey. A bespoke questionnaire consisting of 18 items with varying response formats measuring treatment satisfaction. Items are not combined into a unitary measure.
Number of Materials Accessed | Collects engagement from time of consent to 3-month follow-up
  The system collects information on the number of lessons completed and number of additional resources accessed.
Number of Contacts with Therapist | Collects engagement from time of consent to 3-month follow-up.
  The system collects information on the number of emails and/or phone calls sent to and received from the assigned therapist.
Demographics | Screening
  Demographic questions will be collected at screening for descriptive purposes. No scores are calculated.
Sleep history & treatment history | Screening
  Sleep and treatment history questions will be administered at screening for descriptive purposes. No scores are calculated based on these questions.

CONTACTS AND LOCATIONS:
Overall Officials: Heather D Hadjistavropoulos, PhD, Principal Investigator — University of Regina
Locations (1):
- University of Regina, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Additional information about the PSP Sleep Course. — https://www.pspnet.ca/en/for-psp/online-courses/therapist-guided-psp-sleep-course